CLINICAL TRIAL: NCT02315131
Title: A 2-Stage, Single-Dose Study in Healthy Volunteers and COPD Patients With an Open Label Ipratropium Bromide Reference to Evaluate the Efficacy, Pharmacokinetics, and Safety Profile of Inhaled TV46017
Brief Title: Study in Healthy Volunteers and COPD Patients to Evaluate the Efficacy and Safety of Inhaled TV46017
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TV46017-COPD-10046
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- TV46017- Healthy Volunteers (Experimental): Stage 1 includes a single-dose treatment period
  Interventions: Drug: TV46017
- Placebo - Healthy Volunteers (Placebo Comparator): Some healthy subjects will be randomized to receive placebo.
  Interventions: Drug: Placebo
- TV46017 15 μg- COPD (Experimental): Stage 2 includes two 24 hour treatment periods with approximately 7 days of washout in between each treatment period; and open label ipratropium bromide pressurized metered-dose inhaler hydrofluoroalkane (HFA) will be administered
  Interventions: Drug: TV46017
- TV46017 60 μg- COPD (Experimental): Stage 2
  Interventions: Drug: TV46017
- TV46017 120 μg- COPD (Experimental): Stage 2
  Interventions: Drug: TV46017
- TV46017 240 μg- COPD (Experimental): Stage 2
  Interventions: Drug: TV46017

INTERVENTIONS:
Drug: TV46017 — TV46017 15, 60, 120, and 240 μg; 4 ascending doses of inhaled TV46017 with an ipratropium bromide reference to evaluate the single administration of 4 ascending doses of inhaled TV46017 in COPD patients.
  Other Names: 46017
  Arms: TV46017 120 μg- COPD; TV46017 15 μg- COPD; TV46017 240 μg- COPD; TV46017 60 μg- COPD; TV46017- Healthy Volunteers
Drug: Placebo — Placebo Comparator
  Other Names: Matching placebo
  Arms: Placebo - Healthy Volunteers

SUMMARY:
The primary objective of the study is to characterize the safety profile and duration of bronchodilation of a single dose of inhaled TV46017

ELIGIBILITY:
Stage 1 Inclusion Criteria (healthy volunteers):

* The subject is a male or female 20 to 75 years of age, inclusive, weighing 50 to 80 kg with a body mass index (BMI) of less than 30 kg/m2. Note: Every effort should be made to enroll approximately equal numbers of men and women in each group.
* The subject is in good health as determined by medical and psychiatric history, physical examination, electrocardiogram (ECG), serum chemistry, hematology, urinalysis, and serology.
* Other criteria apply, please contact the investigator for more information

Stage 2 Inclusion Criteria (COPD patients):

* Current or former cigarette smokers with a history of cigarette smoking of ≥10 pack years at the SV (number of cigarette packs smoked per day multiplied by the number of years smoked; eg, 2 packs/day for 3 years equals a 6 pack year history).
* Diagnosis of COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease guidelines.
* Male or female; 40 to 75 years of age, inclusive.
* Patient is free of any other medical conditions or concomitant treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the study.
* Other criteria apply, please contact the investigator for more information

Stage 1 Exclusion Criteria (healthy volunteers):

* History or current evidence of a clinically significant or uncontrolled disease.
* Any disorder that may interfere with the absorption, distribution, metabolism or excretion of study drugs.
* History of severe allergy to milk protein.
* Active smokers or former smokers who quit within 3 months of the first dose of study drug. Former smokers with greater than five-pack years (ie, the equivalent of one pack per day for five years) are also excluded.
* Other criteria apply, please contact the investigator for more information

Stage 2 Exclusion Criteria (COPD patients):

* Recent history of hospitalization due to an exacerbation of airway disease within 3 months.
* Need for increased treatments of COPD within 6 weeks prior to the SV.
* Occurrence of a COPD exacerbation, which is not resolved by 4 weeks or more prior to the SV/informed consent. (Note: An exacerbation of COPD is defined as any worsening of the patient's baseline COPD symptoms requiring any treatment other than rescue albuterol or the patient's regular maintenance therapy. This includes requiring the use of systemic corticosteroids, antibiotics, and/or emergency room visit or hospitalization.)
* History of and/or current diagnosis of asthma.
* Known α1 antitrypsin deficiency, active lung infections (such as tuberculosis or pneumonia), and lung cancer are absolute exclusionary conditions. A patient who, in the opinion of the investigator, has any other significant respiratory condition in addition to COPD should be excluded. Examples may include clinically significant noncystic bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Allergic rhinitis is not exclusionary.
* Other criteria apply, please contact the investigator for more information

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-12h | Baseline, 12 hours
  baseline adjusted forced expiratory volume in 1 second area under the curve over 12 hours

SECONDARY OUTCOMES:
FEV1 | Baseline, 12 hours
  baseline adjusted trough 12 hour
Percentage of Participants with Adverse Events | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (7):
- United States (2):
  - Teva Investigational Site 13033, St Louis, Missouri
  - Teva Investigational Site 13034, Raleigh, North Carolina
- Australia (2):
  - Teva Investigational Site 78984, Adelaide
  - Teva Investigational Site 78985, Nedlands
- New Zealand (3):
  - Teva Investigational Site 79037, Auckland
  - Teva Investigational Site 79036, Hamilton
  - Teva Investigational Site 79034, Wellington